CLINICAL TRIAL: NCT07106203
Title: The Effect of Pursed-Lip Breathing on Physiological Parameters and Discharge Readiness in Children Diagnosed With Pneumonia: A Randomized Controlled Study
Brief Title: Effect of Pursed-Lip Breathing on Physiological Parameters and Discharge Readiness in Children With Pneumonia
Acronym: PLB-PEDPNEU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATU-PLB-2025; B.30.2.ATA.0.01.00/647 (Other: Ataturk Univ Non-Interventional Ethics Committee)
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Pneumonia
Keywords: Pursed-Lip Breathing; Pediatric Pneumonia; Respiratory Function; Discharge Readiness; Physiological Parameters; Pulmonary Rehabilitation; Non-pharmacological intervention
MeSH Terms: conditions — Pneumonia; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This randomized controlled study includes two arms: an intervention group receiving Pursed-Lip Breathing (PLB) exercises twice daily and a control group receiving standard care. The intervention will be performed over a 3-day period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participant group assignments to minimize detection bias. Data analysis will also be conducted by an independent researcher who is unaware of group allocations. Due to the nature of the intervention, participants and intervention providers cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Children aged 3-4 years diagnosed with pneumonia will receive only standard hospital care. No additional respiratory exercise will be applied. Physiological parameters will be measured at the same intervals as the intervention group for comparison.
- PLB Intervention Group (Experimental): Children aged 3-4 years diagnosed with pneumonia will receive Pursed-Lip Breathing (PLB) exercises under nurse supervision, twice daily for three consecutive days. PLB will be performed using playful methods with a toy (e.g., saxophone ball). Respiratory rate, heart rate, and oxygen saturation will be measured before and after each session.
  Interventions: Behavioral: Pursed-Lip Breathing (PLB)

INTERVENTIONS:
Behavioral: Pursed-Lip Breathing (PLB) — Children in the intervention group will receive Pursed-Lip Breathing exercises twice daily for three days under nurse supervision. Exercises will be applied using playful techniques with a toy (e.g., saxophone ball). Physiological parameters will be measured before and after each session.
  Arms: PLB Intervention Group

SUMMARY:
This study aims to evaluate the effects of Pursed-Lip Breathing (PLB) exercises on physiological parameters (such as respiratory rate, heart rate, and oxygen saturation) and discharge readiness in children diagnosed with pneumonia. The study is designed as a randomized controlled trial involving pediatric patients between the ages of 3 and 4. The intervention includes guided PLB exercises performed twice daily for three consecutive days. Data will be collected before and after each session to assess changes in physiological measures and readiness for hospital discharge.

DETAILED DESCRIPTION:
Pneumonia remains one of the leading causes of hospitalization and morbidity in early childhood, often requiring supportive respiratory interventions. Pursed-Lip Breathing (PLB) is a simple, non-pharmacological respiratory technique that has shown promise in improving respiratory function by increasing exhalation time, enhancing oxygenation, and reducing respiratory workload.

This randomized controlled trial aims to evaluate the effects of PLB exercises on physiological parameters (respiratory rate, heart rate, and oxygen saturation) and readiness for hospital discharge in children aged 3-4 years diagnosed with community-acquired pneumonia. Participants will be randomized into intervention and control groups. The intervention group will receive PLB exercises using a toy-based blowing device (saxophone ball blower) twice daily for three consecutive days under supervision, while the control group will receive standard care.

Physiological parameters will be measured immediately before and after each PLB session using standardized methods. In addition, parental perception of discharge readiness will be assessed using the Pediatric Readiness for Hospital Discharge Scale - Parent Form (Ped-RHDS) on the first and third days of hospitalization.

The study hypothesizes that PLB exercises will lead to improved oxygen saturation, reduced respiratory and heart rates, and increased readiness for discharge in the intervention group compared to controls. This research will contribute to the evidence supporting non-pharmacological nursing interventions that can enhance respiratory outcomes and discharge processes in pediatric pneumonia patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 4 years
* Diagnosed with community-acquired pneumonia (CAP), defined as pneumonia occurring in a previously healthy child within 14 days of symptom onset and requiring hospitalization
* The child's primary caregiver is the mother
* Both mother and child must remain in the hospital for at least 3 days
* Hospitalization due to pneumonia with an expected average stay of 4-5 days, based on disease severity and clinical condition
* Mother must be present as a caregiver throughout the hospital stay
* Voluntary participation with signed informed consent from the parent or legal guardian

Exclusion Criteria:

* Presence of any chronic disease in addition to pneumonia
* Mother not staying as a caregiver during hospitalization
* Withdrawal of consent by the mother and/or child
* Discharge before 3 days for any reason (e.g., refusal of treatment, early discharge request)

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Respiratory Rate | Before and after each PLB session over a 3-day intervention period
  Respiratory rate will be measured before and after each PLB session to evaluate the intervention's effect on pulmonary function.
Change in Heart Rate | Before and after each PLB session over a 3-day intervention period
  Heart rate will be recorded before and after each PLB session to assess changes in cardiovascular response.
Change in Oxygen Saturation (SpO₂) | Before and after each PLB session over a 3-day intervention period
  Peripheral oxygen saturation (SpO₂) will be evaluated before and after each PLB session to determine its impact on oxygenation.

SECONDARY OUTCOMES:
Change in Pediatric Readiness for Hospital Discharge Scale - Parent Form (Ped-RHDS) Scores | Day 1 (morning) and Day 3 (evening)
  The Pediatric Readiness for Hospital Discharge Scale - Parent Form (Ped-RHDS) will be administered to parents by an independent nurse on Day 1 (morning) and Day 3 (evening) of hospitalization. The scale evaluates parents' perceptions of their child's readiness for discharge. The total score ranges from 0 to 100, with higher scores indicating a greater perceived readiness for hospital discharge. This outcome measure will be used to assess the effect of the PLB intervention on discharge preparedness.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan KADIROĞLU, Asst Prof, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University Health Sciences Institute and Research Hospital - Department of Pediatrics, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study (after de-identification) will be shared with qualified researchers. Data will be available for secondary analysis upon request, starting 6 months after publication and for a period of 2 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication and ending 2 years later.
Access Criteria: With researchers who submit a methodologically sound proposal and receive approval from the study team.
URL: https://www.beu.edu.tr/personel/e.dursun@beu.edu.tr/iletisim

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT07106203/SAP_000.pdf